CLINICAL TRIAL: NCT04122625
Title: A Dose-optimization, Exploratory Phase Ib/II Study to Assess Safety and Efficacy of the Second Mitochondrial-derived Activator of Caspases (SMAC) Mimetic Debio 1143, When Given in Combination With the Anti-PD-1 Antibody Nivolumab in Patients With Specific Solid Tumors Who Have Progressed During or Immediately After Anti-PD-1/PD-L1 Treatment
Brief Title: Study to Assess Safety and Efficacy of the Second Mitochondrial-derived Activator of Caspases (SMAC) Mimetic Debio 1143
Acronym: SMARTPLUS-106
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1143-106; 2018-003546-16 (EudraCT Number)
Record Dates: First submitted 2019-08-30; First posted 2019-10-10 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A - Debio 1143 150 mg + Nivolumab (Experimental): Participants received Debio 1143, 150 milligrams (mg) capsules, orally once on Days 1 to 10 and Days 15 to 24 of each 28-day treatment cycle along with nivolumab 240 mg, intravenous (IV) infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
  Interventions: Drug: Debio 1143; Drug: Nivolumab
- Part A - Debio 1143 200 mg + Nivolumab (Experimental): Participants received Debio 1143, 200 mg capsules, orally once on Days 1 to 10 and Days 15 to 24 of each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
  Interventions: Drug: Debio 1143; Drug: Nivolumab
- Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab (Experimental): Participants with small-cell lung cancer (SCLC) received Debio 1143, 200 mg capsules, orally once on Days 1 to 28 in each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
  Interventions: Drug: Debio 1143; Drug: Nivolumab
- Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab (Experimental): Participants with squamous cell carcinoma of the head and neck (SCCHN) received Debio 1143, 200 mg capsules, orally once on Days 1 to 28 in each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
  Interventions: Drug: Debio 1143; Drug: Nivolumab
- Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab (Experimental): Participants with gastrointestinal (GI) cancers received Debio 1143, 200 mg capsules, orally once on Days 1 to 28 in each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
  Interventions: Drug: Debio 1143; Drug: Nivolumab
- Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab (Experimental): Participants with gynecologic cancers received Debio 1143, 200 mg capsules, orally once on Days 1 to 28 in each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
  Interventions: Drug: Debio 1143; Drug: Nivolumab

INTERVENTIONS:
Drug: Debio 1143 — Administered as capsules.
Drug: Nivolumab — Administered as IV infusion.

SUMMARY:
Part A (dose-optimization)- to determine the recommended phase 2 dose (RP2D) taking into account dose-limiting toxicity (DLT/s) in Cycle 1, overall safety/tolerability and pharmacokinetic (PK), by optimizing doses of Debio 1143 when combined with the standard dose of nivolumab, as well as treatment compliance in participants with advanced solid malignancies who failed prior systemic standard treatments.

Part B (basket trial)- to evaluate the preliminary anti-tumor activity of Debio 1143 at the RP2D in combination with nivolumab at the standard dose, overall and in each participant cohort (Cohort 1: small cell lung cancer [SCLC]; Cohort 2: squamous cell carcinoma of the head and neck [SCCHN]; Cohort 3: gastrointestinal (GI) cancers with known microsatellite instability-high/mismatch repair deficiency (MSI-H/MMRd) or other deoxyribonucleic acid (DNA) damage repair (DDR) abnormalities, including homologous recombination deficiency (HRD); Cohort 4: platinum-resistant epithelial ovarian cancer [EOC], endometrial cancer, primary peritoneal cancer (PPC) or cervical cancer, with known MSIH/MMRd, hereditary/somatic mutations of the breast cancer 1 (BRCA1) and BRCA2 genes or other DNA DDR abnormalities (incl. HRD).

ELIGIBILITY:
Inclusion Criteria:

* Have received at least one prior line of standard systemic chemotherapy in the advanced/unresectable cancer setting (standard adjuvant/neoadjuvant treatment is acceptable if relapse occurred within six months of treatment end)
* Have progressed or relapsed during or after a prior anti-programmed cell death-1 (PD-1)/ programmed cell death-ligand 1 (PD-L1)-based treatment, given either as a single agent or in combination with standard/approved chemotherapy, tyrosine kinase inhibitors (TKIs), radiotherapy (RT) or other monoclonal antibodies (mAbs) that are not known to modulate/inhibit immune checkpoints (CPIs)
* Measurable disease (Part B only) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or Gynecologic Cancer Intergroup (GCIG) criteria in Cohort #4 of Part B (if applicable) and documented PD during or after prior PD-1/PD-L1 based therapy

Exclusion Criteria:

* Thoracic or head and neck radiation >30 gray (Gy) within the 3 months prior to Cycle 1 Day 1 (C1D1)
* Have received, in total, more than 3 (i.e., Cohorts 1 & 2) or 4 (i.e., Cohorts 3 & 4) lines of prior systemic treatments in Part B (including adjuvant or neoadjuvant regimens if relapse within six months prior to C1D1)
* Liver cirrhosis Child-Pugh score B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber/Partners Cancer Care, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Montefiore Medical Center PRIME, The Bronx, New York
  - UC Health, LLC., Cincinnati, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Methodist Hospital, Houston Methodist Cancer Center, Houston, Texas
  - Georgetown University - Lombardi Comprehensive Cancer Center, Northwest, Washington
- France (3):
  - Centre Leon Berard, Lyon
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - START Madrid, Fundacion Jimenez Diaz, Madrid
  - START Madrid, H.U. Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 24 investigational sites in the United States, Spain, and France from 26 April 2019 to 6 April 2022.
Pre-assignment Details: A total of 46 participants were enrolled in this study, 11 participants with advanced solid malignancies who failed prior systemic standard treatments into Part A and 35 participants into Part B of the study. Part B of the study was started after recommended phase 2 dose (RP2D) was determined in Part A and did not include any participants from Part A.
Period: Part A (up to 2.92 Years)
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Started | 3 | 8 | 0 | 0 | 0 | 0
Completed (Completed also includes 1 participant in arm group, Part A: Debio 1143 200 mg + Nivolumab who entered and completed the extension phase of Part A.) | 1 | 4 | 0 | 0 | 0 | 0
Not Completed | 2 | 4 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 4 | 0 | 0 | 0 | 0
Period: Part B (up to 2.33 Years)
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Started | 0 | 0 | 8 | 8 | 8 | 11
Completed | 0 | 0 | 2 | 0 | 0 | 4
Not Completed | 0 | 0 | 6 | 8 | 8 | 7
Not completed — Patient lost to follow-up | 0 | 0 | 1 | 1 | 2 | 0
Not completed — Death | 0 | 0 | 5 | 7 | 6 | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Groups:
- Part A - Debio 1143 150 mg + Nivolumab: Participants received Debio 1143, 150 mg capsules, orally once on Days 1 to 10 and Days 15 to 24 of each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
- Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab: Participants with SCLC received Debio 1143, 200 mg capsules, orally once on Days 1 to 28 in each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
- Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab: Participants with SCCHN received Debio 1143, 200 mg capsules, orally once on Days 1 to 28 in each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
- Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab: Participants with GI cancers received Debio 1143, 200 mg capsules, orally once on Days 1 to 28 in each 28-day treatment cycle along with nivolumab 240 mg, IV infusion on Days 1 and 15 of each 28-day treatment cycle allowed for a maximum of 26 cycles.
- Total: Total of all reporting groups
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab | Total
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11 | 46
Age, Continuous [Mean (Full Range); unit: years] | 71.0 [58 to 79] | 55.5 [27 to 81] | 65.5 [57 to 74] | 61.6 [48 to 71] | 63.9 [36 to 81] | 64.8 [43 to 79] | 63.0 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 1 | 3 | 11 | 21
  Male | 2 | 7 | 4 | 7 | 5 | 0 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 7 | 5 | 6 | 7 | 6 | 34
  Unknown or Not Reported | 0 | 1 | 2 | 2 | 1 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 7 | 6 | 5 | 7 | 6 | 34
  Race: Other | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: Unknown | 0 | 1 | 2 | 2 | 1 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT: any of following treatment-emergent adverse events (TEAEs) as per NCI CTCAE Grade V5.0 Criteria (Grades 1=mild, 2=moderate, 3=severe and 4 or 5= life-threatening/fatal outcomes) which are possibly, probably or definitely related to combination treatment and occurring in Cycle 1 (1 Cycle=28 days): Any Grade 4 or 5 hematologic toxicity, clinical or laboratory non-hematologic toxicity; febrile neutropenia any grade, Grade 3 thrombocytopenia if associated with bleeding or requiring platelet transfusion; Grade 2; Grade 3 and any other Grade 3 non-hematologic, treatment-related clinical toxicity lasting ≥3 days; delay of >2 weeks due to drug-related toxicity in initiating Cycle 2; unable to complete at least 70% of the scheduled treatment (>six Debio 1143 skipped doses in Cycle 1) due to treatment-related toxicity; required dose reduction in Cycle 1 or on Cycle 2 Day 1 or requirement for treatment withdrawal due to treatment-related toxicity (even if not meeting other DLT criteria).
Time Frame: Part A: Cycle 1 (28 days)
Population: Recommended phase 2 dose (RP2D) population included participants who received at least 70% of Debio 1143 (i.e., a maximum of 6 missed Debio 1143 doses) and at least one nivolumab dose as planned in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Primary Outcome: Part B: Confirmed Objective Response Rate (ORR)
Description: ORR was determined per response evaluation criteria in solid tumors (RECIST) v1.1 and/or gynecologic cancer intergroup (GCIG) criteria (for Cohort 4). ORR was calculated as the percentage of participants with a confirmed objective response. A confirmed objective response is a confirmed best overall response of partial response (PR) or complete response (CR) recorded after the start of study treatment until disease progression/recurrence was documented, a new systemic anti-cancer therapy was started or analysis cut-off, whichever occurred first. CR is defined by the disappearance of all target lesions and reduction of any pathological lymph nodes in short axis to <10 millimeters (mm). PR is defined by at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter.
Time Frame: Part B: From the start of study treatment until disease progression/recurrence was documented, a new systemic anti-cancer therapy was started or analysis cut-off, whichever occurred first (up to approximately 2.05 years)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 8 | 8 | 8 | 11
percentage of participants | 0.0 [0 to 37] | 0.0 [0 to 37] | 0.0 [0 to 37] | 9.1 [0 to 41]

3. Secondary Outcome: Parts A and B: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Including Laboratory Abnormalities Reported as TEAEs, and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial participant administered a medicinal product that does not necessarily have a causal relationship with this treatment. A TEAE is any new, related or non-related, undesirable medical occurrence or change of an existing condition in a participant that occurs during the treatment-emergent period, starting or worsening on or after the first study drug administration and up to 5 months after last nivolumab infusion, or the earliest date of new anticancer therapy - 1 day, whichever occurs first. An SAE is defined as any untoward medical occurrence that at any dose results in death; is life-threatening (i.e., puts the participant at immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect, or is otherwise medically significant.
Time Frame: From the first study drug administration and up to 5 months after last nivolumab infusion, or the earliest date of new anticancer therapy -1 day, whichever occurs first (up to approximately 2.08 years in Part A and 2.05 years in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
Participants
  TEAEs | 3 | 8 | 8 | 8 | 8 | 11
  SAEs | 0 | 8 | 0 | 6 | 5 | 5

4. Secondary Outcome: Parts A and B: Change From Baseline in Weight
Time Frame: From Baseline up to end of treatment (up to approximately 1.53 years in Part A and up to 1 year in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug. Overall number of participants analyzed indicates the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 4 | 7 | 3 | 4 | 8
kilograms (kg) | -5.57 (5.705) | -10.00 (9.416) | -4.33 (3.888) | -4.00 (6.557) | -0.80 (5.415) | -1.11 (1.680)

5. Secondary Outcome: Parts A and B: Number of Participants With Markedly Abnormal Change From Baseline in Vital Signs
Description: Vital sign parameters assessed comprise of systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate. Markedly abnormal criteria for vital signs include SBP [millimeters of mercury (mmHg)]: ≤ 90 mmHg OR change from baseline ≤ -20 mmHg, ≥ 140 mmHg OR change from baseline ≥ 20 mmHg; DBP (mmHg): ≤ 60 mmHg OR change from baseline ≤ -20 mmHg, ≥ 90 mmHg OR change from baseline ≥ 20 mmHg; Heart rate [beats per minute (bpm)]: ≤ 50 bpm OR change from baseline ≤ -20 bpm, ≥ 100 bpm OR change from baseline ≥ 20 bpm.
Time Frame: From Baseline up to end of treatment (up to approximately 1.53 years in Part A and up to 1 year in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Parts A and B: Number of Participants With Change From Baseline in Temperature Reported as TEAEs
Description: Change from baseline in temperature reported as TEAEs included pyrexia. A TEAE is any new, related or non-related, undesirable medical occurrence or change of an existing condition in a participant that occurs during the treatment-emergent period, starting or worsening on or after the first study drug administration and up to 5 months after last nivolumab infusion, or the earliest date of new anticancer therapy - 1 day, whichever occurs first.
Time Frame: From Baseline up to end of treatment (up to approximately 1.53 years in Part A and up to 1 year in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
Participants | 0 | 2 | 1 | 1 | 0 | 3

7. Secondary Outcome: Parts A and B: Number of Participants With Markedly Abnormal Change From Baseline in Electrocardiogram (ECG) Readings
Description: ECG parameters comprised of PR Interval [millisecond (msec)], QRS Interval (msec), QT Interval (msec), QTcB Interval (msec), QTcF Interval (msec), heart rate (HR) (bpm), RR interval (msec), derived HR (msec), calculated as 60000/RR interval [for data checking only: should be within 5% of HR]. Marked abnormal criteria for ECG parameters included absolute values QRS interval: < 50 msec, > 110 msec; absolute values for QT interval, QTcB interval: >450 msec, > 480 msec, > 500 msec, QTcF: > 480 msec, > 500 msec; change from baseline values for QTcB interval, and QTcF: >30 msec increase from baseline, >60 msec increase from baseline. Data for highest on-treatment change from baseline as per the markedly abnormal criteria for ECG parameters are reported. On-treatment is the period of time between the first and last administration of any study drug. Participants with at least one markedly abnormal change from baseline value in the above categories are reported.
Time Frame: From Baseline up to end of treatment (up to approximately 1.53 years in Part A and up to 1 year in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug. Overall number of participants analyzed indicates the number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 2 | 8 | 8 | 8 | 8 | 11
Participants
  QRS duration: >110 msec | 0 | 3 | 1 | 1 | 2 | 0
  QT Interval: >450 msec | 0 | 1 | 2 | 1 | 3 | 0
  QT Interval: >480 msec | 0 | 1 | 0 | 0 | 0 | 0
  QTcB Interval: >450 msec | 2 | 2 | 3 | 5 | 1 | 5
  QTcB Interval: >480 msec | 0 | 0 | 0 | 0 | 1 | 1
  QTcB Interval: >500 msec | 0 | 1 | 0 | 1 | 0 | 0
  QTcB Interval: >30 msec increase from baseline | 0 | 4 | 3 | 5 | 3 | 6
  QTcB Interval: >60 msec increase from baseline | 0 | 0 | 0 | 1 | 0 | 0
  QTcB Interval: >30 msec or >60 msec increase from baseline | 0 | 4 | 3 | 6 | 3 | 6
  QTcF Interval: >480 msec | 0 | 1 | 0 | 0 | 0 | 0
  QTcF Interval: >500 msec | 0 | 0 | 0 | 1 | 0 | 0
  QTcF Interval: >30 msec increase from baseline | 0 | 1 | 2 | 3 | 1 | 4
  QTcF Interval: >60 msec increase from baseline | 0 | 0 | 0 | 1 | 0 | 0

8. Secondary Outcome: Parts A and B: Number of Participants With Shift From Baseline to Worst On-Treatment Value in Eastern Cooperative Oncology Group Performance Status (ECOG-PS)
Description: The ECOG-PS was used to assess the effect of disease progression on participants' daily activities. ECOG-PS is graded as follows: Grade 0 - fully active, able to carry on all pre-disease performance without restriction; Grade 1 - restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; Grade 2 - ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50% of waking hours; Grade 3 - capable of only limited self-care, confined to bed or chair for more than 50% of waking hours; Grade 4 - completely disabled, cannot carry on any self-care, totally confined to bed or chair; Grade 5 - dead. Shift values from baseline grade to worst on-treatment grade and missing values were reported.
Time Frame: From Baseline up to end of treatment (up to approximately 1.53 years in Part A and up to 1 year in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
Participants
  Shift From Grade 0 to Grade 0 | 1 | 3 | 0 | 2 | 1 | 1
  Shift From Grade 0 to Grade 1 | 0 | 2 | 3 | 0 | 2 | 4
  Shift From Grade 0 to Grade 2 | 0 | 1 | 2 | 0 | 1 | 0
  Shift From Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 1 | 0
  Shift From Grade 1 to Grade 1 | 2 | 1 | 2 | 3 | 2 | 5
  Shift From Grade 1 to Grade 2 | 0 | 1 | 1 | 1 | 1 | 0
  Shift From Grade 1 to Grade 3 | 0 | 0 | 0 | 2 | 0 | 0
  Missing | 0 | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Parts A and B: Number of Participants With TEAEs Including Laboratory Abnormalities Leading to Treatment Discontinuations and Dose Modifications
Time Frame: as for outcome 3
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
Participants
  TEAEs Leading to Discontinuation of Debio 1143 | 1 | 1 | 0 | 3 | 1 | 2
  TEAEs Leading to Discontinuation of Nivolumab | 1 | 1 | 0 | 3 | 1 | 2
  TEAEs Leading to Dose Modification of Debio 1143 | 2 | 5 | 5 | 5 | 3 | 4
  TEAEs Leading to Dose Modification of Nivolumab | 2 | 6 | 4 | 5 | 1 | 4

10. Secondary Outcome: Part A: Confirmed Objective Response Rate (ORR)
Description: ORR was determined per RECIST v1.1. ORR was calculated as the percentage of participants with a confirmed objective response. A confirmed objective response is a confirmed best overall response of PR or CR recorded after the start of study treatment until disease progression/recurrence was documented, a new systemic anti-cancer therapy was started or analysis cut-off, whichever occurred first. CR is defined by the disappearance of all target lesions and reduction of any pathological lymph nodes in short axis to <10 mm. PR is defined by at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter.
Time Frame: Part A: From the start of study treatment until disease progression/recurrence was documented, a new systemic anti-cancer therapy was started or analysis cut-off, whichever occurred first (up to approximately 2.08 years)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8
percentage of participants | 0.0 | 12.5

11. Secondary Outcome: Parts A and B: Unconfirmed Objective Response Rate (uORR)
Description: uORR was calculated as the percentage of participants with unconfirmed objective response per RECIST v1.1. Unconfirmed objective response is an unconfirmed best overall response of PR or CR. Objective response was derived as any PR or CR recorded after the start of study treatment until disease progression/recurrence was documented, a new systemic anti-cancer therapy was started or analysis cut-off, whichever occurred first. CR is defined by the disappearance of all target lesions and reduction of any pathological lymph nodes in short axis to <10 mm. PR is defined by at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter.
Time Frame: From the start of study treatment until disease progression/recurrence was documented, a new systemic anti-cancer therapy was started or analysis cut-off, whichever occurred first (up to approximately 2.08 years in Part A and 2.05 years in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
percentage of participants | 0.0 | 25.0 | 0.0 | 0.0 | 0.0 | 9.1

12. Secondary Outcome: Parts A and B: Disease Control Rate (DCR)
Description: DCR was calculated as the percentage of participants with disease control. Disease control was derived as any CR, PR, or stable disease reported during the study. CR is defined by the disappearance of all target lesions and reduction of any pathological lymph nodes in short axis to <10 mm. PR is defined by at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter.
Time Frame: as for outcome 11
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
percentage of participants | 66.7 | 50.0 | 25.0 | 75.0 | 37.5 | 45.5

13. Secondary Outcome: Parts A and B: Median Duration of Response (DOR)
Description: DOR is defined as the time, in months, between date of the initial response (PR or CR) or date of first reduction of 50% in carbohydrate antigen 125 (CA-125), and date of the first documented disease progression or death due to any cause, whichever occurs first. CR is defined by the disappearance of all target lesions and reduction of any pathological lymph nodes in short axis to <10 mm. PR is defined by at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter. Data is reported as Kaplan-Meier product-limit estimates.
Time Frame: as for outcome 11
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug. Overall number of participants analyzed indicates censored participants with at least a CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 1
months |  | NA [NA to NA] — The median and the 95% confidence interval (CI) were not estimable due to insufficient number of participants with events. |  |  |  | NA [NA to NA] — The median and the 95% confidence interval (CI) were not estimable due to insufficient number of participants with events.

14. Secondary Outcome: Parts A and B: Progression Free Survival (PFS)
Description: PFS duration is defined as the time, in months, elapsed between treatment initiation and tumor progression or death from any cause, whichever occurs first.
Time Frame: From the start of study treatment until disease progression/recurrence or death from any cause, whichever occurs first (up to approximately 2.08 years in Part A and 2.05 years in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
months | 2.3 [1.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 2.3 [0.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.8 [1.0 to 3.2] | 1.9 [0.9 to 3.5] | 1.2 [0.8 to 4.2] | 1.8 [1.3 to 5.2]

15. Secondary Outcome: Parts A and B: PFS Rate at Months 6 and 12
Description: PFS is defined as duration elapsed between treatment initiation and tumor progression or death from any cause, whichever occurs first. Data for PFS rate is reported as Kaplan-Meier product-limit estimates and includes Brookmeyer-Crowley confidence intervals.
Time Frame: Months 6 and 12
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug. Number analyzed indicates the number of participants analyzed at the given time points. No participants were analyzed at Month 12 in Part B.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
proportion of participants
  Month 6 | 0.0 [0.0 to 0.0] | 0.2 [0.0 to 0.5] | 0.1 [0.0 to 0.4] | 0.0 [0.0 to 0.0] | 0.1 [0.0 to 0.4] | 0.2 [0.0 to 0.4]
  Month 12: number analyzed (Participants) | 3 | 8 | 0 | 0 | 0 | 0
  Month 12 | 0.0 [0.0 to 0.0] | 0.2 [0.0 to 0.5] |  |  |  |

16. Secondary Outcome: Parts A and B: Overall Survival (OS)
Description: OS is defined as the time elapsed, in months, between treatment initiation and death from any cause.
Time Frame: From the start of study treatment until death from any cause, whichever occurs first (up to approximately 2.08 years in Part A and 2.05 years in Part B)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
months | 13.8 [12.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [1.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 17.5 [3.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 4.7 [0.9 to 13.4] | 5.2 [1.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 11.7 [3.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events.

17. Secondary Outcome: Parts A and B: OS Rate at Months 12 and 18
Description: OS is defined as the time elapsed, in months, between treatment initiation and death from any cause. Data for OS rate is reported as Kaplan-Meier product-limit estimates and includes Brookmeyer-Crowley confidence intervals.
Time Frame: Months 12 and 18
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug. Number analyzed indicates the number of participants analyzed at the given time points.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8 | 8 | 8 | 8 | 11
proportion of participants
  Month 12 | 1.0 [1.0 to 1.0] | 0.5 [0.2 to 0.8] | 0.9 [0.4 to 1.0] | 0.3 [0.0 to 0.6] | 0.4 [0.1 to 0.7] | 0.4 [0.1 to 0.7]
  Month 18: number analyzed (Participants) | 1 | 1 | 8 | 8 | 8 | 11
  Month 18 | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with events. | 0.5 [0.2 to 0.8] | 0.1 [0.0 to 0.4] | 0.4 [0.1 to 0.7] | 0.3 [0.0 to 0.6]

18. Secondary Outcome: Part A: Area Under the Curve From Time 0 to 4 Hours (AUC0-4H) of Debio 1143 and Debio 1143-MET1
Time Frame: Cycle 1: predose, 0.5, 1.5, 4 hours post-dose on Days 1 and 15, predose, 1.5, 4 hours post-dose on Days 8 and 22; Cycle 3: predose, 0.5, 1.5, 4 hours post-dose on Day 1 and predose, 1.5, 4 hours post-dose on Day 15 (each cycle=28 days)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug. Number analyzed indicates the number of participants with available data for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8
hours*nanograms per milliliter (h*ng/mL)
  Debio 1143: Cycle 1 Day 1 | 6200.28 (330.246) | 4907.15 (2496.914)
  Debio 1143: Cycle 1 Day 8: number analyzed (Participants) | 3 | 7
  Debio 1143: Cycle 1 Day 8 | 4321.40 (1127.611) | 5861.53 (3764.659)
  Debio 1143: Cycle 1 Day 15: number analyzed (Participants) | 3 | 7
  Debio 1143: Cycle 1 Day 15 | 5081.21 (868.905) | 5114.03 (3168.408)
  Debio 1143: Cycle 1 Day 22: number analyzed (Participants) | 3 | 5
  Debio 1143: Cycle 1 Day 22 | 4517.00 (3539.938) | 4086.09 (2516.921)
  Debio 1143: Cycle 3 Day 1: number analyzed (Participants) | 3 | 5
  Debio 1143: Cycle 3 Day 1 | 4053.97 (3005.430) | 6844.02 (4940.667)
  Debio 1143: Cycle 3 Day 15: number analyzed (Participants) | 2 | 4
  Debio 1143: Cycle 3 Day 15 | 4725.37 (2033.252) | 5934.72 (2251.520)
  Debio 1143-MET1: Cycle 1 Day 1 | 2624.48 (953.275) | 1662.25 (957.856)
  Debio 1143-MET1: Cycle 1 Day 8: number analyzed (Participants) | 3 | 7
  Debio 1143-MET1: Cycle 1 Day 8 | 3884.59 (565.589) | 5133.24 (3794.465)
  Debio 1143-MET1: Cycle 1 Day 15: number analyzed (Participants) | 3 | 7
  Debio 1143-MET1: Cycle 1 Day 15 | 2104.06 (325.456) | 1673.48 (986.138)
  Debio 1143-MET1: Cycle 1 Day 22: number analyzed (Participants) | 3 | 5
  Debio 1143-MET1: Cycle 1 Day 22 | 3634.33 (1591.770) | 5064.61 (4242.170)
  Debio 1143-MET1: Cycle 3 Day 1: number analyzed (Participants) | 3 | 5
  Debio 1143-MET1: Cycle 3 Day 1 | 983.62 (501.515) | 2617.59 (2250.993)
  Debio 1143-MET1: Cycle 3 Day 15: number analyzed (Participants) | 2 | 4
  Debio 1143-MET1: Cycle 3 Day 15 | 3255.14 (513.699) | 2208.80 (775.572)

19. Secondary Outcome: Part B: AUC0-4H of Debio 1143 and Debio 1143-MET1
Time Frame: Cycle 1: predose, 1.5, 4 hours post-dose on Days 1 and 22; Cycle 3: predose, 1.5, 4 hours post-dose on Day 1 (each cycle = 28 days)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug. Overall number of participants analyzed indicates number of participants available for analysis. Number analyzed indicates the number of participants with available data for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 7 | 7 | 8 | 10
h*ng/mL
  Debio 1143: Cycle 1 Day 1 | 6842.88 (3251.994) | 5552.70 (4559.658) | 5149.10 (1922.588) | 7619.75 (3287.399)
  Debio 1143: Cycle 1 Day 22: number analyzed (Participants) | 7 | 6 | 5 | 8
  Debio 1143: Cycle 1 Day 22 | 7167.67 (4161.553) | 5668.59 (3536.016) | 3218.09 (1137.952) | 6801.02 (1841.871)
  Debio 1143: Cycle 3 Day 1: number analyzed (Participants) | 2 | 2 | 3 | 7
  Debio 1143: Cycle 3 Day 1 | 5674.83 (757.917) | 3248.39 (3165.907) | 2117.23 (970.849) | 5920.77 (2206.953)
  Debio 1143-MET1: Cycle 1 Day 1: number analyzed (Participants) | 7 | 5 | 8 | 10
  Debio 1143-MET1: Cycle 1 Day 1 | 2737.56 (1280.628) | 3440.08 (2274.864) | 2255.49 (1153.863) | 3140.29 (1139.965)
  Debio 1143-MET1: Cycle 1 Day 22: number analyzed (Participants) | 7 | 6 | 5 | 8
  Debio 1143-MET1: Cycle 1 Day 22 | 5938.44 (2187.477) | 10100.42 (3889.091) | 5404.44 (4032.522) | 7085.47 (5196.199)
  Debio 1143-MET1: Cycle 3 Day 1: number analyzed (Participants) | 2 | 2 | 3 | 7
  Debio 1143-MET1: Cycle 3 Day 1 | 3409.44 (2059.973) | 1587.21 (1838.618) | 2381.90 (2767.733) | 2128.83 (1581.498)

20. Secondary Outcome: Part A: Area Under the Curve From Time 0 to 8 Hours (AUC0-8H) of Debio 1143 and Debio 1143-MET1
Time Frame: Cycle 1: predose, 0.5, 1.5, 4, 8 hours post-dose on Days 1 and 15, and predose, 1.5, 4, 8 hours post-dose on Day 8; Cycle 3: predose, 0.5, 1.5, 4, 8 hours post-dose on Day 1 and predose, 1.5, 4, 8 hours post-dose on Day 15 (each cycle = 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 7
h*ng/mL
  Debio 1143: Cycle 1 Day 1 | 8954.45 (1347.640) | 8497.84 (3213.996)
  Debio 1143: Cycle 1 Day 8 | 6699.18 (1315.190) | 9437.55 (6036.801)
  Debio 1143: Cycle 1 Day 15 | 7280.65 (945.078) | 8024.00 (5036.125)
  Debio 1143: Cycle 3 Day 1: number analyzed (Participants) | 2 | 4
  Debio 1143: Cycle 3 Day 1 | 4623.23 (2089.994) | 10627.09 (6520.082)
  Debio 1143: Cycle 3 Day 15: number analyzed (Participants) | 2 | 4
  Debio 1143: Cycle 3 Day 15 | 6864.95 (1815.779) | 9072.05 (3529.268)
  Debio 1143-MET1: Cycle 1 Day 1 | 5940.42 (2217.500) | 5128.38 (2307.490)
  Debio 1143-MET1: Cycle 1 Day 8 | 7743.38 (1258.029) | 10646.90 (8177.450)
  Debio 1143-MET1: Cycle 1 Day 15 | 4921.26 (741.691) | 4304.95 (2105.077)
  Debio 1143-MET1: Cycle 3 Day 1: number analyzed (Participants) | 2 | 4
  Debio 1143-MET1: Cycle 3 Day 1 | 2315.46 (1568.487) | 6632.52 (6610.503)
  Debio 1143-MET1: Cycle 3 Day 15: number analyzed (Participants) | 2 | 4
  Debio 1143-MET1: Cycle 3 Day 15 | 6011.84 (429.313) | 6225.18 (2315.768)

21. Secondary Outcome: Part A: Maximum Observed Concentration (Cmax) of Debio 1143 and Debio 1143-MET1
Time Frame: Cycle 1: Predose,0.5,1.5,4,8 hours post-dose (Days 1 and 15), predose,1.5,4,8 hours post-dose (Day 8), predose,1.5,4 hours post-dose (Day 22); Cycle 3: predose,0.5,1.5,4,8 hours post-dose (Day 1), predose,1.5,4,8 hours post-dose (Day 15) (Cycle=28 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 8
nanograms per milliliter (ng/mL)
  Debio 1143: Cycle 1 Day 1 | 3063.33 (771.838) | 2020.63 (1015.945)
  Debio 1143: Cycle 1 Day 8: number analyzed (Participants) | 3 | 7
  Debio 1143: Cycle 1 Day 8 | 1656.67 (568.624) | 2132.71 (1346.859)
  Debio 1143: Cycle 1 Day 15: number analyzed (Participants) | 3 | 7
  Debio 1143: Cycle 1 Day 15 | 2426.67 (567.656) | 1956.29 (1137.771)
  Debio 1143: Cycle 1 Day 22: number analyzed (Participants) | 3 | 5
  Debio 1143: Cycle 1 Day 22 | 2037.00 (1637.415) | 1528.96 (910.236)
  Debio 1143: Cycle 3 Day 1: number analyzed (Participants) | 3 | 5
  Debio 1143: Cycle 3 Day 1 | 1954.00 (1119.459) | 3071.00 (1928.848)
  Debio 1143: Cycle 3 Day 15: number analyzed (Participants) | 2 | 4
  Debio 1143: Cycle 3 Day 15 | 1970.00 (1244.508) | 2265.00 (886.397)
  Debio 1143-MET1: Cycle 1 Day 1 | 989.67 (344.515) | 972.50 (489.140)
  Debio 1143-MET1: Cycle 1 Day 8: number analyzed (Participants) | 3 | 7
  Debio 1143-MET1: Cycle 1 Day 8 | 1193.33 (222.336) | 1733.23 (1184.636)
  Debio 1143-MET1: Cycle 1 Day 15: number analyzed (Participants) | 3 | 7
  Debio 1143-MET1: Cycle 1 Day 15 | 868.00 (117.051) | 915.86 (390.840)
  Debio 1143-MET1: Cycle 1 Day 22: number analyzed (Participants) | 3 | 5
  Debio 1143-MET1: Cycle 1 Day 22 | 1088.33 (581.758) | 1658.68 (1339.093)
  Debio 1143-MET1: Cycle 3 Day 1: number analyzed (Participants) | 3 | 5
  Debio 1143-MET1: Cycle 3 Day 1 | 611.00 (376.227) | 1343.60 (1078.400)
  Debio 1143-MET1: Cycle 3 Day 15: number analyzed (Participants) | 2 | 4
  Debio 1143-MET1: Cycle 3 Day 15 | 1177.00 (272.943) | 1148.50 (458.398)

22. Secondary Outcome: Part B: Cmax of Debio 1143 and Debio 1143-MET1
Time Frame: as for outcome 19
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 8 | 8 | 8 | 11
ng/mL
  Debio 1143: Cycle 1 Day 1 | 2839.5 (1293.43) | 2266.1 (1830.74) | 2331.3 (823.28) | 2850.0 (1413.87)
  Debio 1143: Cycle 1 Day 22: number analyzed (Participants) | 8 | 6 | 5 | 10
  Debio 1143: Cycle 1 Day 22 | 2786.3 (1591.66) | 2065.8 (1205.31) | 1327.0 (416.30) | 2891.0 (860.28)
  Debio 1143: Cycle 3 Day 1: number analyzed (Participants) | 3 | 2 | 3 | 7
  Debio 1143: Cycle 3 Day 1 | 2183.3 (496.42) | 1726.0 (1094.60) | 975.3 (179.70) | 2271.4 (954.80)
  Debio 1143-MET1: Cycle 1 Day 1 | 1077.38 (473.925) | 1070.71 (808.979) | 1190.00 (439.686) | 1320.00 (483.919)
  Debio 1143-MET1: Cycle 1 Day 22: number analyzed (Participants) | 8 | 6 | 5 | 10
  Debio 1143-MET1: Cycle 1 Day 22 | 1888.50 (668.598) | 2886.67 (915.394) | 1782.80 (1074.434) | 2289.10 (1414.128)
  Debio 1143-MET1: Cycle 3 Day 1: number analyzed (Participants) | 3 | 2 | 3 | 7
  Debio 1143-MET1: Cycle 3 Day 1 | 808.67 (748.505) | 738.00 (724.077) | 965.33 (982.152) | 891.29 (488.887)

23. Secondary Outcome: Part A: Trough Concentration (Cmin) of Debio 1143 and Debio 1143-MET1
Time Frame: Cycle 1: predose on Days 3, 8, 15, 17 and 22; Cycle 3: predose on Days 1, 3, 15, 17; Cycle 6: predose on Day 1
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 6
ng/mL
  Debio 1143: Cycle 1 Day 3 | 113.10 (31.892) | 169.50 (120.014)
  Debio 1143: Cycle 1 Day 8 | 118.27 (30.751) | 173.35 (113.797)
  Debio 1143: Cycle 1 Day 15: number analyzed (Participants) | 1 | 5
  Debio 1143: Cycle 1 Day 15 | 7.34 (NA) — The standard deviation cannot be calculated for 1 participant. | 5.22 (2.844)
  Debio 1143: Cycle 1 Day 17 | 99.37 (19.290) | 133.57 (86.239)
  Debio 1143: Cycle 1 Day 22: number analyzed (Participants) | 3 | 5
  Debio 1143: Cycle 1 Day 22 | 83.53 (19.630) | 173.70 (135.079)
  Debio 1143: Cycle 3 Day 1: number analyzed (Participants) | 1 | 2
  Debio 1143: Cycle 3 Day 1 | 10.20 (NA) — The standard deviation cannot be calculated for 1 participant. | 4.72 (0.410)
  Debio 1143: Cycle 3 Day 3: number analyzed (Participants) | 3 | 2
  Debio 1143: Cycle 3 Day 3 | 110.47 (13.808) | 97.20 (37.901)
  Debio 1143: Cycle 3 Day 15: number analyzed (Participants) | 0 | 2
  Debio 1143: Cycle 3 Day 15 |  | 8.71 (6.640)
  Debio 1143: Cycle 3 Day 17: number analyzed (Participants) | 2 | 3
  Debio 1143: Cycle 3 Day 17 | 118.00 (16.971) | 136.37 (81.772)
  Debio 1143: Cycle 6 Day 1: number analyzed (Participants) | 0 | 1
  Debio 1143: Cycle 6 Day 1 |  | 5.31 (NA) — The standard deviation cannot be calculated for 1 participant.
  Debio 1143-MET1: Cycle 1 Day 3 | 453.33 (180.059) | 620.10 (434.376)
  Debio 1143-MET1: Cycle 1 Day 8 | 387.00 (145.812) | 793.65 (953.516)
  Debio 1143-MET1: Cycle 1 Day 15: number analyzed (Participants) | 1 | 3
  Debio 1143-MET1: Cycle 1 Day 15 | 33.30 (NA) — The standard deviation cannot be calculated for 1 participant. | 6.39 (3.241)
  Debio 1143-MET1: Cycle 1 Day 17 | 543.00 (154.182) | 531.93 (560.633)
  Debio 1143-MET1: Cycle 1 Day 22: number analyzed (Participants) | 3 | 5
  Debio 1143-MET1: Cycle 1 Day 22 | 367.33 (289.588) | 805.78 (961.228)
  Debio 1143-MET1: Cycle 3 Day 1: number analyzed (Participants) | 1 | 2
  Debio 1143-MET1: Cycle 3 Day 1 | 6.97 (NA) — The standard deviation cannot be calculated for 1 participant. | 23.65 (27.655)
  Debio 1143-MET1: Cycle 3 Day 3: number analyzed (Participants) | 3 | 2
  Debio 1143-MET1: Cycle 3 Day 3 | 443.67 (172.631) | 1157.50 (1304.612)
  Debio 1143-MET1: Cycle 3 Day 15: number analyzed (Participants) | 0 | 2
  Debio 1143-MET1: Cycle 3 Day 15 |  | 13.55 (9.687)
  Debio 1143-MET1: Cycle 3 Day 17: number analyzed (Participants) | 2 | 3
  Debio 1143-MET1: Cycle 3 Day 17 | 611.00 (322.441) | 639.67 (387.727)
  Debio 1143-MET1: Cycle 6 Day 1: number analyzed (Participants) | 0 | 1
  Debio 1143-MET1: Cycle 6 Day 1 |  | 3.15 (NA) — The standard deviation cannot be calculated for 1 participant.

24. Secondary Outcome: Part B: Trough Concentration (Cmin) of Debio 1143 and Debio 1143-MET1
Time Frame: Cycle 1: predose on Days 8 and 22; Cycle 3: predose on Day 1 (each cycle = 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 8 | 8 | 7 | 10
ng/mL
  Debio 1143: Cycle 1 Day 8: number analyzed (Participants) | 6 | 7 | 7 | 10
  Debio 1143: Cycle 1 Day 8 | 198.05 (143.494) | 167.20 (112.649) | 192.86 (130.457) | 143.39 (44.663)
  Debio 1143: Cycle 1 Day 22: number analyzed (Participants) | 8 | 6 | 5 | 10
  Debio 1143: Cycle 1 Day 22 | 150.29 (80.118) | 221.60 (140.039) | 130.92 (50.555) | 146.39 (50.852)
  Debio 1143: Cycle 3 Day 1: number analyzed (Participants) | 2 | 2 | 2 | 5
  Debio 1143: Cycle 3 Day 1 | 3.24 (0.721) | 11.08 (12.056) | 3.50 (0.318) | 4.94 (2.137)
  Debio 1143-MET: Cycle 1 Day 8: number analyzed (Participants) | 6 | 8 | 7 | 10
  Debio 1143-MET: Cycle 1 Day 8 | 693.33 (983.009) | 1917.89 (1826.669) | 1005.20 (1150.843) | 1118.40 (710.330)
  Debio 1143-MET1: Cycle 1 Day 22: number analyzed (Participants) | 8 | 6 | 5 | 10
  Debio 1143-MET1: Cycle 1 Day 22 | 658.50 (557.846) | 2103.33 (1410.308) | 830.20 (827.444) | 1113.04 (811.962)
  Debio 1143-MET1: Cycle 3 Day 1: number analyzed (Participants) | 2 | 2 | 0 | 3
  Debio 1143-MET1: Cycle 3 Day 1 | 2.84 (0.255) | 14.35 (11.809) |  | 10.30 (3.751)

25. Secondary Outcome: Part A: Serum Trough Concentration of Nivolumab
Time Frame: Cycle 1: predose, 1.5, 8 hours post-dose on Day 15; Cycle 3: predose, 0.5, 1.5, 8 hours post-dose on Day 1 and predose, 1.5 hours post-dose on Day 15 (each cycle = 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 3 | 7
ng/mL
  Cycle 1 Day 15 | 21366.67 (4808.673) | 22271.43 (7553.744)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1
  Cycle 3 Day 1 | 43500.00 (NA) — The standard deviation cannot be calculated for 1 participant. | 32700.00 (NA) — The standard deviation cannot be calculated for 1 participant.
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 1
  Cycle 3 Day 15 |  | 27100.00 (NA) — The standard deviation cannot be calculated for 1 participant.

26. Secondary Outcome: Part B: Serum Trough Concentration of Nivolumab
Time Frame: Cycle 1: predose, 1.5 hours post-dose on Day 15; Cycle 3: predose, 1.5 hours post-dose on Days 1 and Day 15; Cycle 6: predose on Day 1 (each cycle = 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 8 | 7 | 8 | 10
ng/mL
  Cycle 1 Day 15 | 21312.5 (2942.51) | 25414.3 (8766.68) | 33725.0 (17751.28) | 22332.0 (8864.61)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 6
  Cycle 3 Day 1 | 34100.0 (NA) — The standard deviation cannot be calculated for 1 participant. | 40600.0 (NA) — The standard deviation cannot be calculated for 1 participant. |  | 43866.7 (11670.08)
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 1 | 0 | 4
  Cycle 3 Day 15 |  | 45400.0 (NA) — The standard deviation cannot be calculated for 1 participant. |  | 58400.0 (10492.22)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Cycle 6 Day 1 |  | 40400.0 (NA) — The standard deviation cannot be calculated for 1 participant. |  |

27. Secondary Outcome: Parts A and B: Time to Response (TTR)
Description: The average of the time taken in days for PR is reported. PR is defined by at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameter.
Time Frame: as for outcome 11
Population: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug. Overall number of participants analyzed indicates the number of participants with at least a CR or PR.
Measure: Mean (Full Range); unit: days
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
Number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 1
days |  | 82 [56 to 108] |  |  |  | 52 [52 to 52]

ADVERSE EVENTS:
Time Frame: From after the first study drug administration and up to 5 months after last nivolumab infusion, or the earliest date of new anticancer therapy -1 day, whichever occurs first (up to approximately 2.08 years in Part A and 2.05 years in Part B)
Description: Safety analysis set included all participants who were enrolled and received at least one dose of any study drug.
Arm/Group | Part A - Debio 1143 150 mg + Nivolumab | Part A - Debio 1143 200 mg + Nivolumab | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/8 | 5/8 | 7/8 | 6/8 | 7/11
Serious Adverse Events (participants affected / at risk) | 0/3 | 8/8 | 0/8 | 6/8 | 5/8 | 5/11
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 8/8 | 8/8 | 8/8 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Debio 1143 150 mg + Nivolumab (N=3) | Part A - Debio 1143 200 mg + Nivolumab (N=8) | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab (N=8) | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab (N=8) | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab (N=8) | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Debio 1143 150 mg + Nivolumab (N=3) | Part A - Debio 1143 200 mg + Nivolumab (N=8) | Part B - Cohort 1 (SCLC): Debio 1143 200 mg + Nivolumab (N=8) | Part B - Cohort 2 (SCCHN): Debio 1143 200 mg + Nivolumab (N=8) | Part B - Cohort 3 (GI Cancers): Debio 1143 200 mg + Nivolumab (N=8) | Part B - Cohort 4 (Gynecologic Cancers): Debio 1143 200 mg + Nivolumab (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 2 | 2 | 4
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 1 | 6 | 3 | 2 | 2
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 0 | 3
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fungal Foot Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lip Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 1 | 5
Amylase increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 4
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 2 | 2 | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 3 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 4 | 2 | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Listeria encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
VIth nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Cortisol decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or scientific communication related to this study can only take place once the agreement between the Sponsor and the Investigator has been reached.

DOCUMENTS (2):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT04122625/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT04122625/SAP_001.pdf